CLINICAL TRIAL: NCT05502107
Title: A Multicenter, Stepped Wedge, Cluster Randomized Study of a Prehospital Sepsis Protocol and Its Impact on Timely Antibiotic Administration in the Emergency Department and Subsequent Adverse Events
Brief Title: Impact of a Prehospital Sepsis Protocol on Timely Antibiotic Administration and Subsequent Adverse Events
Acronym: IMPRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carmen Polito, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004512; U54CK000601-01-01 (Other Grant/Funding Number: Centers for Disease Control and Prevention (CDC)); U54CK000601-01 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Sepsis
Keywords: Sepsis screening; EMS-based screening
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: This is a multicenter, cluster-randomized, stepped-wedge implementation study of an EMS sepsis screening and early communication protocol. Each study cluster represents one EMS organization and one partnered acute care hospital. Each cluster pair will participate in both a baseline and intervention phase of study varying between 6-18 months each (baseline and intervention), in approximately 6 month blocks, depending on the order of cluster randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRESS Intervention (Experimental): Study sites will participate in the intervention phase for 6 to 18 months, depending on the order of cluster randomization. Sites will switch from the baseline phase in approximately 6 month blocks, with all sites delivering the intervention for the final 6 months of the study.
  Interventions: Behavioral: PRESS Intervention
- Standard of Care (No Intervention): Study sites will participate in the standard of care phase to collect baseline data for 6 to 18 months, depending on the order of cluster randomization. All sites are in the baseline phase for the first 6 months then sites will switch one at a time, every 6 months, to the intervention phase of the study.

INTERVENTIONS:
Behavioral: PRESS Intervention — The study intervention is PRESS protocol training and educational delivered to EMS providers, followed by protocol implementation. EMS providers will be trained to screen all EMS patients for protocol eligibility and will start using the protocol at the beginning of the intervention phase. The PRESS EMS protocol includes 2 major components: 1) an evidence-based sepsis screening tool, and 2) a prehospital sepsis alert call to the receiving hospital for participants who screen positive. Upon arrival to the ED, ED providers will provide immediate medical assessment to the patient to determine whether there is concern for sepsis. If the treating provider determines there is concern for sepsis, the provider will deliver usual sepsis care per local hospital protocols, workflows, or care pathways. Sepsis treatment interventions will not be specified by this study protocol.
  Arms: PRESS Intervention

SUMMARY:
The primary purpose of this study is to evaluate the impact of an Emergency Medical Services (EMS) based sepsis screening and early warning protocol on the timing of early sepsis care in the Emergency Department (ED).

DETAILED DESCRIPTION:
Sepsis is life-threatening medical emergency and a common cause of morbidity and mortality among hospitalized patients. Recognizing and treating sepsis immediately is key to achieving optimal patient outcomes after sepsis. The prehospital, EMS setting represents a unique opportunity to implement best practice by operationalizing guideline-recommended, system-wide sepsis screening protocols in an effort to facilitate earlier recognition of sepsis and minimize delays in evaluation and treatment. Unfortunately, evidence-based screening tools to assist EMS providers in recognizing this heterogenous syndrome are lacking, and recognition by EMS providers is generally poor.

The purpose of this study is to evaluate the prehospital sepsis (PRESS) protocol, which is an evidence-based sepsis screening and early communication protocol designed for use in the prehospital, EMS environment. The PRESS protocol pairs a validated sepsis screening tool with a prehospital sepsis alert to the receiving ED for patients who are screen positive. This innovative approach has been used to improve patient care and outcomes in other life-threatening, time-sensitive medical emergencies including heart attack and stroke. Prehospital screening and an early warning call to the ED before patient arrival provides valuable lead time that makes immediate evaluation and treatment by EMS providers possible once a patient arrives in the ED.

This study includes three study sites which are each comprised of cluster pairs of one EMS organization and one partnered acute care hospital. Each cluster pair will participate in both a baseline and intervention phase of study. EMS providers will be trained to screen for sepsis according to the PRESS protocol. The PRESS EMS protocol includes 2 major components: 1) an evidence-based sepsis screening tool, and 2) a prehospital sepsis alert call to the receiving hospital for participants who screen positive. Upon arrival to the ED, ED providers will provide immediate medical assessment to the patient to determine whether there is concern for sepsis. The overarching hypothesis is that implementation of an EMS-based sepsis screening and early warning protocol will be associated with a reduction in time first antibiotic administration in the ED among patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Lowest EMS systolic blood pressure <110 mmHg
* Highest EMS pulse rate >90 beats per minute
* Highest EMS respiratory rate >20 breaths per minute
* EMS transport to a participating study ED/hospital
* At least one of the following present:

  * Lowest systolic blood pressure <90 mmHg
  * Age 40 years or greater
  * Hot temperature assessment or temp >38 degrees Celsius
  * Oxygen saturation <90%
  * Nursing home patient
  * Emergency Medical Dispatch classification = 'sick person'

Exclusion Criteria:

* Any of the following EMS conditions present:

  * Trauma injury
  * Cardiac arrest
  * Psychiatric emergency
  * Toxic ingestion
  * Pregnant patient
* Inability to administratively link EMS and ED/hospital records
* Patient left emergency department prior to being evaluated by a medical provider (inability to classify sepsis status)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 984 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Time to First Antibiotic Administration in the ED | During ED stay on Day 1
  Among eligible EMS patients with sepsis, the time from ED arrival to first antibiotic administration (parenteral only) in the ED will be examined. Time will be censored at the time of hospital admission or ED discharge.

SECONDARY OUTCOMES:
EMS Documentation of Sepsis | During ED stay on Day 1
  Among eligible EMS patients with sepsis, the proportion with EMS documentation of suspected or possible sepsis or positive PRESS screen will be assessed.
EMS Documentation of a Prehospital Sepsis Alert | During ED stay on Day 1
  Among eligible EMS patients with sepsis, the proportion who receive sepsis bundle care within 3 hours of ED arrival (sepsis bundle = blood culture order, lactic acid order, antibiotic administration) will be assessed. Care bundle elements will be analyzed individually and in composite.
Time to Sepsis Bundle from ED Arrival | During ED stay on Day 1
  Among eligible EMS patients with sepsis, the time to sepsis bundle care elements from ED arrival will be assessed. Time will be censored at the time of hospital admission or ED discharge.
Time to First Care Provider Documentation | During ED stay on Day 1
  Among all eligible EMS patients, the time from ED arrival to first care provider documentation in the ED will be assessed.
Proportion of Patients Without Sepsis Receiving Antibiotics in the ED | During ED stay on Day 1
  Among all eligible EMS patients without sepsis, the proportion who receive antibiotic administration (parenteral only) in the ED will be assessed.
Antibiotic Days of Therapy | Up to 10 days (on average)
  The total number of antibiotic days of therapy (DOT) will be assessed. Antibiotic DOT is measured as last calendar day of consecutive antibiotic therapy minus the first calendar day of antibiotic therapy, among patients with and without sepsis.
Proportion of Patients Admitted to the ICU | During hospital stay (up to 20 days, on average)
  Among all eligible EMS patients with and without sepsis, the proportion admitted from the ED directly to ICU level of care will be assessed, stratified by sepsis status.
Hospital Length of Stay | During hospital stay (up to 20 days, on average)
  Among all eligible EMS patients with and without sepsis, total hospital length of stay will be assessed, stratified by sepsis status. Hospital length of stay is defined as days since ED arrival to day of hospital discharge.
In-hospital Death | During hospital stay (up to 20 days, on average)
  In-hospital death among patients with and without sepsis will be assessed, stratified by sepsis status.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen C Polito, MD, MSc, Principal Investigator — Emory University; Jonathan E Sevransky, MD, MHS, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
A limited, de-identified, participant-level dataset will be shared. This dataset will include participant demographics, EMS physiologic data, as well as sepsis screening, classification, and outcomes data.
Supporting Information: Study Protocol
Time Frame: Data will become available starting after publication of the primary study manuscript (anticipated start date July 2025) and will be available through the Emory Dataverse indefinitely.
Access Criteria: A limited data set will be available to the general public for the purposes of conducting analyses such as a secondary analysis or meta analysis. Data can be accessed through the Emory Dataverse after requesting access from the primary study investigator.

REFERENCES:
- [Derived] Das S, Ahmed A, Capurro O, Carr MJ, Castedo FB, Fridkin SK, Hall A, House S, Kellogg J, Kroll M, Kurtzman N, Manjunath R, Mehta CC, Mohr NM, Prakash-Asrani R, Rudolph CC, Spainhour C, Trehan T, Sevransky JE, Polito CC. Protocol for a multicenter, cluster-randomized, stepped-wedge, implementation trial of a prehospital sepsis protocol. Trials. 2025 Nov 11;26(1):491. doi: 10.1186/s13063-025-09172-3. PMID 41220003